CLINICAL TRIAL: NCT05241561
Title: Open-label, Multicenter, Prospective Phase 2 Study to Evaluate the Duration of Treatment With Cabozantinib Among Patients With Metastatic or Locally Advanced Renal Cell Carcinoma on Hemodialysis (HD).
Brief Title: Cabo-POLARIS : A Trial to Evaluate Cabozantinib Among Haemodialysied Patients
Acronym: Cabo-POLARIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/653
Record Dates: First submitted 2022-01-21; First posted 2022-02-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Cancer of Kidney
MeSH Terms: conditions — Kidney Neoplasms | interventions — cabozantinib; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental)
  Interventions: Drug: Cabozantinib; Biological: Blood sample; Other: Questionnaires of quality of life

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be prescribed following its Marketing Authorization with an initiation at a reduced dose of 40 mg per day. The dose will be adjusted according to safety.
  At the end of the first cycle, patients may be eligible for an increase in the dose of cabozantinib (up to 60 mg per day) if the following criteria are met: no adverse effects of grade 3 or 4 cabozantinib-related, no dose reduction or interruption for safety reasons, no long-lasting grade 2 cabozantinib-related adverse effects requiring maximum supportive care. Continuation to 40 mg per day or reduction to 20 mg per day are the other alternatives depending on the safety profile.
Biological: Blood sample — biomonitoring and pharmacokinetics
Other: Questionnaires of quality of life — FKSI-19 and FKSI-DRS and EUROQOL EQ-5D-5L

SUMMARY:
Among patients with renal cell carcinoma (RCC), 2.7 to 4.7 % of patients are at risk of progressing to dialysis or transplantation after partial and radical nephrectomy respectively. Of note, similar risk factors can be seen in both disease: RCC and renal impairment leading to dialysis. Currently, three types of systemic therapies (ST) are mainly used among patients with metastatic renal cell carcinoma (mRCC): anti-angiogenics (mostly tyrosine kinase inhibitors and bevacizumab), mTOR inhibitors and immune checkpoint inhibitor.

ST prescription for patients undergoing HD may be more dangerous than in other patients. This is partially explained by the fact that several adverse events can be induced by both the ST and HD e.g. thromboembolic disease, or hypertension.

Patients in HD are usually excluded from major clinical trials and available data concerning safety and activity of ST in this specific population are lacking. In most cases, drugs' label is driven by the eligibility criteria of large randomized phase 3 trials that exclude this type of patients. The main source of information for these patients comes from academic publications of patients' cases or small cohorts, but they are not included within the drug label. Moreover, no clear guidelines are given by savant societies regarding those patients.

It is known that patients with HD are at high risk of specific adverse events that can sometimes overlap with the safety profile of anti-cancer drugs: thromboembolic complications, cardio-vascular comorbidities, hematologic and metabolic abnormalities.

Having a dedicated clinical trial to this particular population would definitely help the community to improve the care of HD patients by getting prospective data in order to increase the level of evidence and therefore to optimize anticancer drug use in this specific population.

ELIGIBILITY:
Main Inclusion Criteria:

1. Documented histological diagnosis of advanced or metastatic renal cell cancer with a clear-cell or papillary component.
2. Must have received at least one prior line of systemic therapy.
3. Undergoing haemodialysis for more than 3 months without major complications that might confound the results of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
4. Recovery to baseline or ≤ Grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless AE(s) are considered clinically nonsignificant by the investigator and/or stable on supportive therapy.
5. Age eighteen years or older on the day of consent.
6. Karnofsky Performance Status (KPS) score of ≥ 70%.
7. Adequate organ and marrow function.

Main exclusion Criteria:

1. Prior treatment with cabozantinib.
2. Kidney cancer without clear-cell or papillary component.
3. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before cabozantinib initiation.
4. Receipt of any type of anticancer antibody within 2 weeks before randomization. For investigational antibody the delay is 4 weeks.

5 Major surgery within 4 weeks or major radiotherapy within 2 weeks prior to starting cabozantinib. Previous palliative radiotherapy (≤ 10 fractions) for metastatic lesions is permitted, provided that this has been completed at least 48 hours prior to starting cabozantinib. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.

6. Known brain metastases or spinal compression unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 6 weeks before randomization. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of randomization. Patients with a past history of meningeal carcinomatosis are not eligible.

7. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

7a. Cardiovascular disorders

7b Active infection requiring systemic treatment.

7c. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation

7d. Clinically significant haematuria, hematemesis, or haemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary haemorrhage) within 3 months before randomization.

7e. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.

7f. Lesions invading major pulmonary blood vessels. 7g. Other clinically significant disorders.

8. Corrected QT interval > 480 msec within 1 month before randomization. Three ECGs must be performed. If the average of these three consecutive results for QTcF is ≤ 480 msec, the subject meets eligibility in this regard.

9. - Existence of a past history of cancer within 3 years prior to inclusion into the study (excluding cured localized cancer such as non-melanomatous skin cancers, superficial bladder cancers, or in situ for breast or uterine cervical cancer, and localized prostate cancer without biochemical PSA relapse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
rate of patients permanently discontinuing for any reason cabozantinib at 6 months after initiation of treatment | 6 months

SECONDARY OUTCOMES:
rate of patients permanently discontinuing cabozantinib at 6 months after initiation of treatment due to toxicity | 6 months
progression free survival | 24 months
Absolute and relative frequency of dose reductions and temporary or permanent discontinuation of cabozantinib | 24 months
total duration of treatment with cabozantinib | 24 months
progression-free survival (PFS) | 24 months
overall survival (OS) | 24 months
objective response rate | 24 months
overall safety profile of cabozantinib | 24 months
time to deterioration in quality of life on cabozantinib | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No